CLINICAL TRIAL: NCT03768843
Title: Surgical Outcome of Type II Odontoid Fracture, Harms Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, ahmed salaheldin mohammed saro, Assistant professor of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohag3
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Tramatic Odontoid Fracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- traumatic odontoid fracture (Other): C1 C2 fusion screws
  Interventions: Procedure: Harms technique

INTERVENTIONS:
Procedure: Harms technique — Atlantoaxial fusion
  Other Names: C1 C2 fusion

SUMMARY:
Cervical trauma is a common cause of disability following spinal cord injury, especially in athletic populations. The biomechanics in the atlantoaxial joint carry more than 50% of the rotational movement which can be affected in transverse ligament tear associated with odontoid fracture type II. Odontoid fracture type II considered an unstable fracture with a high rate of non-union in conservative treatment. Limitation of the odontoid screws in some cases gives the chance of posterior cervical fixation to have the superior role. Use of polyaxial screws in Harms technique gives the best results in maintaining the majority of the biomechanics.

Purpose: our aim in this study to evaluate Harms technique in those patients regarding pain improvement and restoration of the motor power and to report the complications.

Study design: A retrospective case series study. We Used the Frankel grading system to evaluate the postoperative neurological state.

DETAILED DESCRIPTION:
After approval of Research Ethics Committee, twelve patients with post-traumatic odontoid fracture type II were scheduled in our Neurosurgery department at Sohag University Hospital for atlantoaxial fusion using polyaxial C1 lateral mass and C2 pedicle screws between January 2015 and January 2018.

ELIGIBILITY:
Inclusion Criteria:

1. C1-C2 displacement that needs intra-operative reduction
2. Short neck not suitable for anterior odontoid screw
3. Osteoporotic patients
4. Odontoid fracture associated with transverse ligament tear suspected.
5. Oblique line of fracture
6. Failure of union after conservative treatment.

Exclusion Criteria:

* Associated spinal fractures
* Other comorbidities

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
evaluation neurological deficit using Frankel grading system within 3 years | 3 years
  grades from A to E and A is the best neurological function while E is the worst neurological function

CONTACTS AND LOCATIONS:
Overall Officials: Hisham A Elsharkawy, Professor, Study Director — Sohag faculty of medicine
Locations (1):
- Ahmed Salaheldin Mohammed Saro, Sohag, Egypt